CLINICAL TRIAL: NCT07110116
Title: Comparison of Effects of Alternate Nostril Breathing Exercise With Incentive Spirometer Technique on Lung Functions Among Asthma Patients
Brief Title: Alternate Nostril Breathing With Incentive Spirometry on Lung Function Among Asthma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/02192 Hira Qazi
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternate nostril breathing with Incentive Spirometery (Experimental)
  Interventions: Other: Alternate nostril breathing with Incentive Spirometery
- Incentive Spirometery (Active Comparator)
  Interventions: Other: Incentive spirometery

INTERVENTIONS:
Other: Alternate nostril breathing with Incentive Spirometery — Participants in experimental group were instructed to close their left nostril by left index finger and inhale through their right nostril for six seconds, then closing the right nostril and holding breath for six seconds. Afterward, they exhaled through the left nostril slowly for six seconds. Next, they inhaled through left nostril, keeping the right nostril closed for six seconds then hold the breath by closing both nostrils for six seconds subsequently, and then exhaled through the right nostril, keeping the left closed for six seconds repeating these steps several times for 10 minutes
  Arms: Alternate nostril breathing with Incentive Spirometery
Other: Incentive spirometery — The control group participants were asked to do breathing exercise with incentive spirometry. The subject is asked to create a tight seal around the mouthpiece and asked to inhale deeply and slowly and the subject would observe the flow meter for visual feedback of his/her effort. At the end of the inspiration the subject is asked to sustain the inhalation 2-3 seconds to facilitate the Inspiratory hold. Subject relaxes the seal around the mouthpiece and exhales. Normal breathing is taken, then the exhalation phase in the incentive spirometry is done and the whole cycle is repeated 5 - 10 times thrice a day over a period 6 weeks
  Arms: Incentive Spirometery

SUMMARY:
To compare effects of Alternate Nostril Breathing exercise with incentive spirometer on lung functions (forced vital capacity, forced expiratory volume, and peak expiratory flow rate) in Asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed male & female asthma patients of age 18-60 years.
* Patients with mild to moderate asthma having predicted FEV1 between 60-80%.
* Stable asthma condition without recent exacerbations.
* Able to perform spirometry and follow instructions for the interventions.
* No recent respiratory infections.

Exclusion Criteria:

* Patients with severe asthma (FEV1 < 60% predicted).
* Patients having respiratory infections, recent exacerbations or other comorbidities.
* Inability to perform breathing exercises or spirometry.
* Patients using medications like oral steroids, beta blockers.
* Pregnant women due to potential risks with breathing exercises.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second | 6 week
  Forced Expiratory Volume in 1 second (FEV1) is a measurement of how much air a person can forcefully exhale from their lungs in one second
Forced Vital Capicity | 6 week
  Forced vital capacity (FVC) is a measurement of lung function that quantifies the maximum amount of air a person can forcefully exhale after taking the deepest breath possible
Peak Expiratory Flow Rate | 6 week
  Peak expiratory flow rate (PEFR) measures the maximum speed of air that a person can forcefully exhale in one breath
Asthama Control Test | 6 week
  The Asthma Control Test (ACT) is scored by assigning a value from 1 to 5 to each response in the 5-question survey, then summing these values for a total score ranging from 5 to 25. A higher score indicates better asthma control. A score of 20 or higher generally suggests well-controlled asthma.
Asthama Quality of Life Questionaire with standardized Activities | 6 week
  The Standardized Asthma Quality of Life Questionnaire (AQLQ(S)) is a 32-item questionnaire used to assess the impact of asthma on an individual's quality of life, specifically focusing on the physical, emotional, and social aspects. 7-point Likert scale (7 = not impaired at all - 1 = severely impaired). Scores range 1-7, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Allied Specialist Hospital & Clinics, Abbottābād, Khyber PkahtoonKhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No